CLINICAL TRIAL: NCT03499431
Title: Longitudinal Registry of Endovascular Thoracoabdominal Aneurysms: Study of Fenestrated and Branched Stent Grafts in the Treatment of Aortic Aneurysms
Brief Title: Longitudinal Registry of Endovascular Thoracoabdominal Aneurysms
Acronym: LoRETA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tara Mastracci (Other)
Collaborators: University Hospital, Lille (Other); Skane University Hospital (Other)
Responsible Party: Sponsor-Investigator, Tara Mastracci, Co-Investigator, Royal Free Hospital NHS Foundation Trust
Organization: Royal Free Hospital NHS Foundation Trust (Other)
Other Study IDs: 001
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Aneurysm; Aortic Aneurysm
MeSH Terms: conditions — Aneurysm; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular Thoracoabdominal Aneurysm Repair — Standard of care, treatment of thoracoabdominal aneurysms using endovascular techiniques.
  Other Names: Branched and Fenestrated Devices

SUMMARY:
The purpose of this study is to evaluate the long-term safety and performance of complex endovascular aneurysm repair by inclusion in a longitudinal registry

DETAILED DESCRIPTION:
This is a Global, multicenter, prospective, observational, non-randomized, single-arm, open clinical study will evaluate the long term (i.e. >5 years) safety and efficacy of complex endovascular repair

This study will enroll all patients treated with Fenestrated and Branched devices in Europe and Canada that follow all inclusion criteria and none of the exclusion criteria. The total duration of the study will be of approximately 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility for enrolment shall be based on known information at the time of the procedure. Information obtained at a later date may contradict these criteria, but this will not be considered a deviation of the Study Plan.

Inclusion criteria

A patient is deemed suitable for inclusion in the study if the patient meets both of the following criteria:

1. Patient requires endovascular repair of a thoracic, thoraco-abdominal or abdominal aortic or aorto-iliac aneurysm having morphology suitable for endovascular repair with complex endograft.
2. Patients (or their legal representative for minor patients) who do not object to (oral non-objection declaration, and signed consent form) collection and transmission of his/her data.

Exclusion Criteria:

* Patients are excluded from enrolment into the study if any of the following are true:

  1. Patients whose imaging follow-up is impossible, i.e. patients who are not able to send their follow up CT scans or Duplex US

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing complex EVAR at study sites.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-30 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Longterm Aneurysm Related Mortality | 7 years
  Death attributed to aneurysm rupture